CLINICAL TRIAL: NCT01849237
Title: Russian Single-center Open Randomized Clinical Trial of the Impact of Mesenchymal Stromal Cells Therapy on Organ Dysfunction and 28-day Mortality in Patients With Septic Shock and Severe Neutropenia.
Brief Title: Russian Clinical Trial of Mesenchymal Cells in Patients With Septic Shock and Severe Neutropenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, MD PhD, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuMCeSS
Record Dates: First submitted 2013-05-01; First posted 2013-05-08 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Septic Shock; Nonchemotherapy Drug-induced Neutropenia; Neutropenia After Chemotherapy in Oncohematological Patients; Neutropenia in Patients With Aplastic Anemia
Keywords: Mesenchymal Stromal Cells; Septic Shock; Neutropenia; Procalcitonin; Interleukin-6; Interleukin-10; C-reactive protein; Survival; Organ dysfunction
MeSH Terms: conditions — Shock, Septic; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy of septic shock (Active Comparator): according to Surviving Sepsis Campaign 2012 Antibiotic therapy Fluid therapy Vasopressors Inotropic therapy Steroids
  Interventions: Drug: Standard therapy of septic shock
- Mesenchymal stromal cells+ standard therapy of septic shock (Experimental): MSCs intravenous infusion of 1-2 millions/kg/day will be performed not more than 10 hs after onset of septic shock in patients with severe neutropenia(≤ 1x10^9/l).
  according to Surviving Sepsis Campaign 2012: Antibiotic therapy Fluid therapy Vasopressors Inotropic therapy Steroids
  Interventions: Genetic: Mesenchymal stromal cells; Drug: Standard therapy of septic shock

INTERVENTIONS:
Genetic: Mesenchymal stromal cells — MSCs intravenous infusion of 1-2 millions/kg/day will be performed not more than 10 hs after onset of septic shock in patients with severe neutropenia(≤ 1x10^9/l).
  Arms: Mesenchymal stromal cells+ standard therapy of septic shock
Drug: Standard therapy of septic shock — Antibiotic therapy Fluid therapy Vasopressors Inotropic therapy Steroids

SUMMARY:
Septic shock remains a significant clinical problem associated with high rates of mortality among neutropenic patient despite antimicrobial therapy and supportive care. Recently, mesenchymal stromal cells (MSC) have demonstrated remarkable potential effect in sepsis. MSC treatment significantly reduced mortality in septic mice receiving appropriate antimicrobial therapy. MSCs reduced systemic inflammatory cytokine levels in mice, down-regulated of inflammation and inflammation-related genes (such as interleukin-10, interleukin-6). Bacterial clearance was greater in MSC-treated mice. Thus, MSCs have beneficial effects on experimental sepsis and suggest that MSСs-therapy may be an effective adjunctive treatment to reduce sepsis-related mortality.

The safety of MSCs is proved by Graft-versus-host disease treatment MSCs in patients after bone marrow transplantation.

This study hypothesis is that MSCs reduce organ dysfunction/injury, systemic inflammation and mortality in patients with septic shock and severe neutropenia.

The main goal of the study is to evaluate the impact of MSCs therapy on organ dysfunction/injury, systemic inflammation and 28-day mortality in patients with septic shock and severe neutropenia. All patients will be randomized in two groups: control group (standard treatment of septic shock) and MSCs-group (standard treatment of septic shock + MSCs infusion of 1-2 millions/kg/ day).

DETAILED DESCRIPTION:
All activities related to this human subjects research have been guided by ethical principles and have been reviewed and approved Federalwide Assurance National Ctr for Hematology, FWA00006482. The goal of the trial is to evaluate plasma concentration of proinflammatory cytokine interleukin-6 and the antiinflammatory cytokine interleukin-10, plasma levels of blood creatinine, bilirubin, procalcitonin, C-reactive protein. Then we will evaluate requirement for renal replacement therapy, requirement for mechanical ventilation or non-invasive mechanical ventilation, pulmonary function-coefficient, partial oxygen pressure arterial blood level, electrocardiograms, Kaplan - Meier curve,28-days mortality.

ELIGIBILITY:
Inclusion Criteria:

septic shock

≤10 hs after onset of septic shock severe neutropenia(≤ 1 10^9/l) Patients ≥17 years Signed Informed Consent to treatment

Exclusion Criteria:

oncohematological patients with resistance to chemotherapy Unsigned Informed Consent to treatment Age >75 years; Pregnancy

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days

SECONDARY OUTCOMES:
Evaluation of MSC therapy effects on organ dysfunction | At Baseline and at day 2,3,7,14,21,28
  1. Liver: levels of serum total bilirubin, transaminases, lactate dehydrogenase, plasma protrombin level
  2. Pancreas: amylase level
  3. Renal: number of hemodialysis/ hemodiafiltration, blood urea and creatinine levels
  4. Pulmonary: requirement for mechanical ventilation or non-invasive mechanical ventilation, pulmonary function-coefficient, partial oxygen pressure arterial blood level
  5. Cardiac: requirement for vasopressors, main parameters obtained from Transpulmonary Thermodilution- Systemic Vascular Resistance Index ( SVRI ), Cardiac Output (CO)
Evaluation of MSC therapy effects on systemic inflammatory parameters | At Baseline and at day 2,3,7,14,21,28
  plasma concentration of proinflammatory cytokine IL-6 and the antiinflammatory cytokine IL-10, concentration of procalcitonin, C-reactive protein Fibrinogen level, lactate level , the factor XII-dependent fibrinolytic activity blood routine examination
Evaluation of MSC therapy effects on septic shock reversal | At Baseline and at day 2,3,7,14,21,28
  SOFA score

CONTACTS AND LOCATIONS:
Overall Officials: Gennady M. Galstyan, MD PhD, Principal Investigator — National Research center of Hematology
Locations (1):
- National Research Center for Hematology, Moscow, Russia

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Mei SH, Haitsma JJ, Dos Santos CC, Deng Y, Lai PF, Slutsky AS, Liles WC, Stewart DJ. Mesenchymal stem cells reduce inflammation while enhancing bacterial clearance and improving survival in sepsis. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1047-57. doi: 10.1164/rccm.201001-0010OC. Epub 2010 Jun 17. PMID 20558630
- [Background] Kebriaei P, Robinson S. Treatment of graft-versus-host-disease with mesenchymal stromal cells. Cytotherapy. 2011 Mar;13(3):262-8. doi: 10.3109/14653249.2010.549688. Epub 2011 Jan 13. PMID 21231805